CLINICAL TRIAL: NCT03055429
Title: Enhancing Care of the Aged and Dying in Prisons Phase II
Brief Title: Enhancing Care of the Aged and Dying in Prisons Ph II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Penn State University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0314; 2R42AG049570-02 (NIH)
Record Dates: First submitted 2016-12-13; First posted 2017-02-16 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Aging Problems
Keywords: Prisoners; End-of-life care; Geriatric care; Palliative care; Hospice care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full Scale Unit (Experimental): Testing of 6 modules
  Interventions: Other: Full Scale Unit

INTERVENTIONS:
Other: Full Scale Unit — Pre-test, usability, post-test

SUMMARY:
The mission of corrections is to provide custody, control and care for incarcerated individuals. United States prisons are required by constitutional law to provide adequate care for growing numbers of older inmates who will likely spend their final days in prison. This Phase II project focuses on the correct users accessing correct learning strategies in the correct setting (i.e., interdisciplinary prison staff accessing high quality products designed to educate and lead practice change initiatives within the walls of prisons), by continuing research and development of a learning system that promotes an integrated systems approach to enhancing the care of the aged and dying in prisons.

DETAILED DESCRIPTION:
The United States has the highest rate of incarceration in the world. There are over 1,821 state and federal prisons housing over 2.3 million prisoners in the United States. The demographics of the prison population are shifting. Longer sentences and constrained options for early release compound this trend. The older adult segment of prison populations has more than tripled since 1990. The health status of aging inmates does not mirror the free-world population. In fact, prisoners typically present with health issues common to free citizens who are 10-15 years their senior. Prisoners are wards of that state, that is, the system is responsible for providing for not only custody and control of offenders, but also their care. Collectively, these trends have had a profound impact on prison systems: U.S. prisons are facing sharply increased demands in caring for aged and dying inmates. In response to this need, Phase I project Enhancing Care for the Aged and Dying in Prisons (ECAD-P) demonstrated that (1) there is a need and interest for products such as ECAD-P (i.e., corrections administrators and staff are interested in end-of-life (EOL) care training); (2) trainings should be short, intensive, engaging, interactive, and contextually sensitive to the specific environment; and (3) an interactive, media-rich prototype with high acceptability and usability could be developed. The specification document and commercialization plan indicate it is possible to develop a full-scale ECAD-P learning system in Phase II and market potential exists. The technological innovation proposed for the ECAD-P project is well-suited to the targeted market. Technical merit, feasibility, and market potential of the ECAD-P Learning System were demonstrated in the Phase I project. The purpose of this Phase II application is to continue research and development of the ECAD-P learning system with an emphasis on developing a scalable unit for commercialization and testing scale-up in a larger number of more diverse contexts. More specifically, the aims of ECAD-P Phase II are to 1) Develop a full scale media-rich interactive computer-based learning system consisting of six modules addressing EOL and geriatric care issues in prisons; 2) Conduct in-person usability testing of the full scale ECAD-P Learning System in state and federal prisons to evaluate the user interface, ease of use, and perceived barriers in order to optimize the scalable unit for broader dissemination; and 3) Test scale-up of the full scale ECAD-P Learning System in 12 federal (n=6) and state (n=6) prisons across the nation to evaluate outcomes, usage patterns, and commercialization opportunities. Continued research and development will permit the refinement the scalable unit for commercialization. Expanded testing of the learning system will establish the effectiveness of the learning system and will provide critical insights relevant to dissemination of the commercial product.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Employed by a participating state or federal prison
* Able to speak English
* Able to consent

Exclusion Criteria:

* Under 18 years
* Not employed by a participating state or federal prison
* Unable to speak English
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change of knowledge from Baseline (pre-test) to post-test (4-months). (End-of-Life and geriatric-related knowledge) | Pre-test and Post-test (4-months)
  A questionnaire will be developed using the content expertise of study personnel and consultants. The questionnaire will evaluate the change in knowledge of geriatric-related and end-of-life prior to the training (pre-test) and at the end of the training (post-test @ 4 months)

SECONDARY OUTCOMES:
Environmental Survey via questionnaire | 6 months
  Evaluation of support systems and prison environment.
Environmental Survey via Qualitative Interviews | 6 months
  Evaluation of support systems and prison environment.
Survey of past users of the Toolkit for Enhancing End-of-Life Care in Prisons | 6 months
  Explore the experiences of early adopters of the original Toolkit.
System Usability Questionnaire | 6 months
  The System Usability Scale (SUS) is a validated tool for assessing the usability and acceptability of technology-based products

CONTACTS AND LOCATIONS:
Overall Officials: Janice Penrod, PhD, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - Klein Buendel, Inc., Golden, Colorado
  - Penn State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner P, Sakala L. Mass incarceration: the whole pie. Northampton, MA: Prison Policy Initiative. Available at: Retrieved from: http://www.prisonpolicy.org/reports/pie.html. Published 2014. Updated.
- [Background] Williams BA, Goodwin JS, Baillargeon J, Ahalt C, Walter LC. Addressing the aging crisis in U.S. criminal justice health care. J Am Geriatr Soc. 2012 Jun;60(6):1150-6. doi: 10.1111/j.1532-5415.2012.03962.x. Epub 2012 May 29. PMID 22642489
- [Background] Aday RH. Aging prisoners : crisis in American corrections. Westport, Conn.: Praeger; 2003.